CLINICAL TRIAL: NCT00725218
Title: Phase IV Study of Flurbiprofen Axetil for Uterine Contraction Pain After Abortion
Brief Title: Flurbiprofen Axetil for Uterine Contraction Pain
Acronym: FAUCOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-MZ203; M089732
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-05

CONDITIONS: Postoperative Pain
Keywords: NSAIDs; Postoperative pain; Analgesia; Abortion
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Sodium Chloride; Ringer's Solution; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Saline 5 ml injection 10 min prior to propofol administration.
  Interventions: Drug: Saline
- 2 (Experimental): Flurbiprofen Axetil 50 mg in 5 ml injection 10min prior to propofol administration.
  Interventions: Drug: Flurbiprofen Axetil

INTERVENTIONS:
Drug: Saline — Saline 5 ml injection 10 min prior to propofol administration.
  Other Names: Ringer's solution
  Arms: 1
Drug: Flurbiprofen Axetil — Flurbiprofen Axetil 50 mg in 5 ml injection 10min prior to propofol administration.
  Other Names: KaiFen
  Arms: 2

SUMMARY:
Uterine contraction pain is a common problem after abortion. Optimal analgesic for such suffering is still needed to be guaranteed. Flurbiprofen Axetil is a target-distributable non-steroidal anti-inflammatory drug (NSAID) functioning via block the synthesis of prostaglandin E (PGE). The investigators hypothesized that Flurbiprofen Axetil could suppress the uterine contraction pain after abortion effectively.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II
* Performing abortion operation (medical- or drug-induced
* Requiring painless abortion

Exclusion Criteria:

* < 19yrs, and >= 45yrs
* History of central active drugs administration
* Drug abuse
* Hypertension
* Diabetes
* Any other chronic diseases
* Allergy to the study drugs
* Habit of over-volume alcohol drinking
* Records of history of centrally active drug use and psychiatry
* Any organic disorders

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
VAS pain scorings | At the end of the operation, 0,5,15,30,60min after operation

SECONDARY OUTCOMES:
Anesthetic consumptions | At the end of the operation
Overall VAS satisfaction scorings with analgesia | At the end of the study
Side effects | During the whole period of the study
Volume of bleeding | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China